CLINICAL TRIAL: NCT02463630
Title: Posterior Compression - Distraction Reduction (CDR) Technique in the Treatment of Basilar Invagination Associated With Atlantoaxial Dislocation
Brief Title: Posterior Compression Distraction Reduction （CDR）Technique in the Treatment of BI-AAD
Acronym: CDR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: The Second Hospital of Hebei Medical University (Other); The First Affiliated Hospital of Zhengzhou University (Other); Southern Medical University, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: PCRT
Record Dates: First submitted 2015-06-01; First posted 2015-06-04 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-01

CONDITIONS: Basilar Invagination Associated With Atlantoaxial Dislocation
Keywords: basilar invagination; atlantoaxial dislocation; surgery; restoration technique

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Compression distraction reduction (Experimental): All the participants in this group will be performed Posterior Compression Distraction Reduction Technique for reduction of basilar invagination and atlantoaxial dislocation
  Interventions: Procedure: Posterior Approach Compression Distraction Reduction

INTERVENTIONS:
Procedure: Posterior Approach Compression Distraction Reduction — Patients was placed in prone position. Via midline skin incision, expose the occipital squama and spinal process, vertebral plate and facet joints of C2. 2 multi-axial screws were inserted into the bilateral C2 or C3 pedicles. The posterior edge of the FM up to the lower boundary of cerebellar tonsil (width, 3mm) was removed. A compression occipital plate (COP) was fixed to the occipital bone. 2 titanium rods connect C2/C3 screws and plate heads bilaterally. The COP screw cap was screwed in, compress the beginning of the pre-bending formed titanium rod downward, driving the odontoid process forward to restore the horizontal dislocation. After restoration of horizontal dislocation is confirmed, applying distraction force between the occipital screw and the C2 pedicle screws, restore the vertical dislocation. tight up the screw cap. Graft bone was harvested from the posterior inferior iliac crest bone and implanted into posterior end of the foramen magnum and posterior lamina of axis.

SUMMARY:
Posterior compression - distraction reduction technique （CDR） in the treatment of Basilar invagination associated with atlantoaxial dislocation

DETAILED DESCRIPTION:
Basilar invagination (BI) refers to the skull base into the direction of cervical spine, mainly to the odontoid process into the foramen magnum is a major change of congenital cranial vertebral junction malformation. Different from trauma or inflammatory lesions, there exists not only in horizontal but also vertical direction dislocation between atlas and axis，At present there is no satisfactory and widely accepted operation method. At present, the main treatment strategy is adopt skull traction to patients preoperative or intraoperative and make vertebra X-ray observation. If the skull traction restored the atlanto-axial dislocation, This case belongs to restorable atlanto-axial dislocation. If the skull traction cannot restore the dislocation, that is non-restorable atlanto-axial dislocation. For the restorable type, posterior occipital cervical internal fixation and fusion should be performed. For the non restorable cases, the main theories is that various ligaments and scars is formed between the anterior arch of atlas and the odontoid process lead to the causes of the longitudinal traction, so transoral anterior atlanto-axial joint lysis is needed first, and then adopt posterior occipital-cervical internal fixation and interbody fusion after the atlanto-axial dislocation is restored. Because the anterior trans-oral atlanto-axial joint lysis has weakness of difficult and high risk, it has limit the popularization of the treatment of atlanto-axial dislocation. Currently only a few several spinal surgery centers have the ability to carry out. Another problem of this treatment strategy is that the function of posterior operation confined to occipital-cervical fixation in situ but not considered the try to adopt the posterior open reduction, this is mainly due to the current clinical application of occipital cervical posterior fixation system be lack of the pressure reduction effect.

Abumi proposed posterior operation incision, atlanto-axial restore intraoperative technique in 1999, and designed the first compression screw that has a restore function in the operation. But it hasn't been widely used because of the intraoperative reposition and internal fixation instrument design is not reasonable and the restore technique has a lot of deficiencies In 2006 Wangchao reported another posterior atlanto-axial dislocation reduction technology. The restore direction of this technology is more reasonable than Abumi's, but the occipital titanium plate adopted in this kind of restore technique is still evolved the occipital-cervical internal fixation system designed by Abumi, just have the mechanical properties of restore level atlanto-axial dislocation. but for atlanto-axial dislocation caused by the Basilar invagination is still need to adopt restore by skull traction. And in many cases also need to perform anterior transoral atlanto-axial joint lysis in order to achieve expected reduction effect.

Wangchao adopt the same occipital-cervical internal fixation system as Abumi technique to perform pressure reduction of atlanto-axial dislocation. This technology is more reasonable in the pressing direction. Using the occipital-cervical internal fixation system was same as Abumi technique it doesn't own the function of Distraction reduction. Therefore for the vertical dislocation of atlanto-axial Still need to restore by skull traction, some patients need the anterior transoral atlanto-axial joint lysis to restore by traction.

In 2010 the members of the project group reported the atlanto-axial dislocation restore by simple posterior screw internal fixation technique and has achieved effect. We can restore vertical dislocation between the atlanto-axial effectively by applying distraction force between occipital screws and axis pedicle screws. For those Basilar Invagination (BI) complicated with Atlanto-axial dislocation(AAD), the rate of Atlanto-axial reduction100% reached 65%. But due to the use of internal fixation system is ordinary occipital cervical internal fixation system （Summit system，DePuy Co) lacking of the function pressure reduction, therefore the effect of level reduction of atlanto-axial dislocation is poor. In some cases it induct atlanto-axial joint rearward opening angle increases(picture 5), odontoid falling backwards aggregately, the medulla spinal cord angle narrowed further[10].Furthermore, Part of the reasons why atlanto occipital complex malformation patients failed to achieve 100% reduction is that atlanto-axial lateral is deformities seriously, utual locking, it is difficulty to restore by this technology.

The technology divided intraoperative reduction process into two operating. First of all, restore the level of dislocation between atlanto-axial through pressure, and then restore the vertical dislocation between atlanto-axial through distraction. I designed the compression occipital plate (COP) owned functions both compression and distraction reduction in order to make it convenient in intraoperative technical operation. This type of titanium plate has been obtained the national patent, Patent certificate No. ZL 201320355786.X. The investigation report of Patent Bureau indicated that the design of this type of titanium plate is creative and novel.

The clinical application of this technique has achieved initial success in the treatment of basilar invagination complicated with atlanto-axial dislocation patients. This technology so far is the most reasonable posterior reduction technology in the treatment of basilar invagination complicated with atlanto-axial dislocation mechanics mechanism.

This type of titanium plate has been obtained the national patent, Patent certificate No. ZL 201320355786.X.

Although the compression distraction reduction technology has obvious advantages analyzed from the mechanical properties of angle application of pressurized occipital titanium plate, but if the application of this technology can be safely effective cure basilar invagination and atlanto-axial dislocation patients, improve neurological function, still need further prospective clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-70
* Patients with cervical CT display that atlanto occipital fusion or partial fusion, Atlantoodontoid interval(ADI)>>3mm, odontoid tip over Qian line(CL)>>3mm.
* Agreed to the surgical operation treatment
* The patient can carry out clinical follow-up and agree to long-term clinical follow-up
* Signed informed consent

Exclusion Criteria:

* Patients with traumatic atlanto-axial dislocation
* Patients with rheumatoid atlantoaxial dislocation
* Patients with a history of occipital cervical junction operation
* Patients with severe cerebellar tonsillar hernia (reach the C2 margin), needed to remove tonsil of cerebellum
* Patients during pregnancy and the postpartum period within 3 months
* The life expectancy of < 1 years
* Severe dementia(MMSE<18)
* Severe renal failure (CR > 2.5mg/dl)
* Serious cardiovascular disease (such as unstable angina, heart failure)
* Atrial fibrillation and other severe arrhythmia
* Without the ability to sign the informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Record the patients' cervical JOA score, ASIA score | three days before surgery
  record the basic information of the patients before operation, to evaluate the
The first follow-up after surgery Record the patients' cervical JOA score, ASIA | 3rd day post operation
  MRI.Performed imaging evaluation by radiology doctors.
ADI, CL and Cervicomedullary angle(CMA) by COP system and Compression Distraction Reduction， (CDR) | 3rd day post operation
  ADI, CL and Cervicomedullary angle(CMA) calculations. All the patients perform posterior compression - distraction reduction, occipitocervical internal fixation and interbody fusion applied by COP system and Compression Distraction Reduction， (CDR)

SECONDARY OUTCOMES:
The second follow-up after operation Record the patients' cervical JOA score, ASIA score | 6 months post operation
  Outpatient review at 6 months after surgery, adopt related neurological

CONTACTS AND LOCATIONS:
Overall Officials: Zan Chen, MD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- BEIJING, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Goel A. Treatment of basilar invagination by atlantoaxial joint distraction and direct lateral mass fixation. J Neurosurg Spine. 2004 Oct;1(3):281-6. doi: 10.3171/spi.2004.1.3.0281. PMID 15478366
- [Result] Behari S, Kalra SK, Kiran Kumar MV, Salunke P, Jaiswal AK, Jain VK. Chiari I malformation associated with atlanto-axial dislocation: focussing on the anterior cervico-medullary compression. Acta Neurochir (Wien). 2007 Jan;149(1):41-50; discussion 50. doi: 10.1007/s00701-006-1047-3. Epub 2006 Nov 27. PMID 17131067
- [Result] Jian FZ, Chen Z, Wrede KH, Samii M, Ling F. Direct posterior reduction and fixation for the treatment of basilar invagination with atlantoaxial dislocation. Neurosurgery. 2010 Apr;66(4):678-87; discussion 687. doi: 10.1227/01.NEU.0000367632.45384.5A. PMID 20305492
- [Result] Wang C, Yan M, Zhou HT, Wang SL, Dang GT. Open reduction of irreducible atlantoaxial dislocation by transoral anterior atlantoaxial release and posterior internal fixation. Spine (Phila Pa 1976). 2006 May 15;31(11):E306-13. doi: 10.1097/01.brs.0000217686.80327.e4. PMID 16688020
- [Result] Abumi K, Takada T, Shono Y, Kaneda K, Fujiya M. Posterior occipitocervical reconstruction using cervical pedicle screws and plate-rod systems. Spine (Phila Pa 1976). 1999 Jul 15;24(14):1425-34. doi: 10.1097/00007632-199907150-00007. PMID 10423787